CLINICAL TRIAL: NCT06637826
Title: Study on the Relationship Between Indoor Environment, Use of Personal Disinfection Products, and Human Health
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Xiang Jianbang, Professor, National Natural Science Foundation of China
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: SYSU_SPHSZ_2024099
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: Quaternary Ammonium Disinfectants; Disinfectants; Indoor Environment; Human Health
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blank Control Group (No Intervention)
- Disinfectant Use Control Group (Experimental)
  Interventions: Behavioral: Quaternary Ammonium Compound Disinfectants; Behavioral: Alcohol-based Disinfectants

INTERVENTIONS:
Behavioral: Quaternary Ammonium Compound Disinfectants — Participants are instructed to use quaternary ammonium compound disinfectants during the 1st month (first intervention) and the 3rd month (second intervention) after enrollment, following the guidelines provided. The products include:
  * Laundry disinfectant: Use at least twice per week.
  * Hand sanitizing wipes: Use at least twice per day, individually packaged, recommended for use before meals.
  * Surface disinfecting wipes: Use at least twice per day, individually packaged or multi-pack, recommended for use on surfaces in dormitories or classroom desks.
  * Floor disinfecting wipes: Use at least twice per week, in multi-pack, recommended for use on the floor in personal activity areas in dormitories. These wipes can be used by hand or foot to wipe the floor.
  After each use of the disinfectant products, participants are required to take a photo and send it to the research team as documentation.
  Arms: Disinfectant Use Control Group
Behavioral: Alcohol-based Disinfectants — Participants are instructed to use alcohol-based disinfectants during the 1st month (first intervention) and the 3rd month (second intervention) after enrollment, following the guidelines provided. The products include:
  * Laundry disinfectant: Use at least twice per week.
  * Hand sanitizing wipes: Use at least twice per day, individually packaged, recommended for use before meals.
  * Surface disinfecting wipes: Use at least twice per day, individually packaged or multi-pack, recommended for use on surfaces in dormitories or classroom desks.
  * Floor disinfecting wipes: Use at least twice per week, in multi-pack, recommended for use on the floor in personal activity areas in dormitories. These wipes can be used by hand or foot to wipe the floor.
  After each use of the disinfectant products, participants are required to take a photo and send it to the research team as documentation.
  Arms: Disinfectant Use Control Group

SUMMARY:
Research Purpose and Significance:

Quaternary ammonium compounds (QACs), as cationic surfactants, are widely used in disinfectants, cosmetics, fabric softeners, hair conditioners, and other personal care products. They are a class of emerging organic pollutants commonly found in various environmental media. Existing studies have shown that QACs exhibit immunotoxicity, reproductive toxicity, and developmental toxicity, which has led to increasing concern in developed countries such as Europe and the United States regarding their potential health risks. In 2015, the U.S. Food and Drug Administration (FDA) required manufacturers to provide more human safety data when adding QACs to personal care products. In 2016, the European Union banned the use of benzalkonium chloride in hand sanitizers and body washes. California, USA, announced that it will prohibit the use of Quaternium-15 in cosmetics and personal care products starting in 2025. Currently, China lacks health risk-based regulatory policies for QACs, highlighting a significant gap compared to developed countries. There is an urgent need to conduct detailed assessments of QAC pollution and human exposure to establish a foundation for evaluating the health risks associated with QACs.

In summary, investigating QAC pollution and human exposure in indoor environments is critical for understanding their health risks and will provide important theoretical support for establishing environmental health standards for QACs in China.

Research Methods:

1. Participant Recruitment:

   This study will adopt a panel study design, recruiting 80 young student volunteers from an existing cohort.
2. Study Design:

   Participants will be randomly assigned to two groups in a randomized crossover trial. Group A will use quaternary ammonium compound (QAC) disinfectant products (including laundry disinfectant, hand sanitizing wipes, and surface and floor disinfecting wipes), while Group B will use alcohol-based disinfectant products, both for a period of one month. After the first intervention, there will be a one-month washout period, followed by a crossover intervention where the groups switch products for another month. Participants will wear a custom environmental monitoring device according to the guidelines and will regularly complete health questionnaires, functional assessments, and biological sample collections.
3. Exposure Measurement:

   External exposure to organic compounds in the environment will be monitored using silicone wristbands, while internal exposure will be assessed using blood and urine samples.
4. Health Indicator Measurement:

   A combination of health scales and biochemical tests will be used to assess related health indicators. Health measurements will be conducted four times-once before and once after each intervention. Each session will include the following: a health questionnaire, 10 mL of fasting blood, 40 mL of morning urine, cognitive tests, EEG tests, near-infrared brain imaging, respiratory metabolic tests, arterial function tests, and body composition tests.
5. Statistical Analysis:

Mixed-effects models and machine learning algorithms will be employed to assess the health effects of QAC and alcohol-based disinfectant products on the human body.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled at Sun Yat-sen University Shenzhen Campus
* Willing to voluntarily participate, able to complete questionnaire surveys, exposure measurements, health scale assessments, and biological sample collection (including blood and urine)

Exclusion Criteria:

* Smoking
* Physically weak, unable to fully participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
64 Participants with Disinfectant Products-Related Adverse Events | From enrollment to the end of treatment at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University, Shenzhen, China